CLINICAL TRIAL: NCT02595411
Title: Reliability of the Melbourne Assessment
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: MA_Reliability_2015
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Cerebral Palsy; Stroke; Traumatic Brain Injury; Meningomyelocele; Central Nervous System Diseases
Keywords: Children; Rehabilitation; Upper Limb; Assessments; Outcome Measures
MeSH Terms: conditions — Cerebral Palsy; Stroke; Brain Injuries, Traumatic; Meningomyelocele; Central Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to investigate the reliability of the Melbourne Assessment.

DETAILED DESCRIPTION:
Children with central motor disorders will be tested twice within one week with the Melbourne Assessment. The assessments will be video scored. At a later time point, different raters will rate the same video for inter-rater reliability, the same rater will score the same video for intra-rater reliability, and the same rater will score the repeated assessment videos for test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

* central motor disorders
* ambulant or stationary patients of the Rehabilitation Center Affoltern am Albis
* ability to understand test instructions
* ability to sit upright for 25 minutes
* minimal activity in the assessed upper limb

Exclusion Criteria:

* severe visual and/or auditory problems
* acute lesion in the to assessed upper limb
* lack of compliance

Ages: 30 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with central motor disorders and impaired upper limb function
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Melbourne Assessment 2 | 2 assessments within 1 week
  Assessment to measure unilateral upper limb function

CONTACTS AND LOCATIONS:
Overall Officials: Hubertus van Hedel, PD Dr., Principal Investigator — University Children's Hospital Zurich, Rehabilitation Centre Affoltern am Albis
Locations (1):
- University Children's Hospital Zurich, Rehabilitation Centre Affoltern am Albis, Affoltern am Albis, Switzerland

IPD SHARING:
Plan to Share IPD: No